## INFORMED CONSENT FORM / CONTROL GROUP

- **Document Date**: 12 June 2023
- **Title of The Study**: The Effect of Acupressure on Fatigue, Quality of Life and Comfort in Hemodialysis Patients. Randomized Controlled Study
- NCT Number: 05892679
- **Document**: Informed Consent Form / Control Group

**NCT Number:** 05892679

The Effect of Acupressure on Fatigue, Quality of Life and Comfort in Hemodialysis Patients. Randomized Controlled Study

## INFORMED CONSENT FORM / CONTROL GROUP

Dear Participant;

I am conducting a research titled "The Effect of Acupressure on Quality of Life, Comfort and Fatigue in Hemodialysis Patients, Randomized Controlled Study" in order to determine the effect of acupressure on quality of life, comfort and fatigue in patients receiving hemodialysis treatment.

I hope you will also participate in this study. Participation in the research is on a voluntary basis. Before your decision, I want to inform you about the research. The information obtained will only be used for research purposes and will not be used for any other purpose. Personal information will not be disclosed in the presentation of the research. Your name will not be used within the scope of your participation in this research and your identity rights will be protected. You will not be charged any fee for participating in this research, and you will not be paid any additional fees for participating. You may refuse to participate in this research. You also have the right to withdraw your consent at any stage of the research. We thank you for your participation and support.

I have read all the explanations in the Informed Consent Form. Written and verbal explanations regarding the above-mentioned research were given to me by the researcher named below. I know that I participated in the research voluntarily and I can leave the research at any time with or without justification. I agree to participate in the research in question voluntarily, without any pressure or coercion.

Date: Date:

Volunteer Participant Interview Witness Name, surname: Name, surname:

Tel:

Signature: Signature:

Date:

Researcher interviewing the participant

Name, surname, title: MSN Nurse, Vecihe DÜZEL GÜNDÜZ

**Tel:** 05056733313

**Signature:** 

NCT Number: 05892679

The Effect of Acupressure on Fatigue, Quality of Life and Comfort in Hemodialysis Patients. Randomized Controlled Study